CLINICAL TRIAL: NCT00809783
Title: A PHASE 3, MULTICENTER, RANDOMIZED, LONG TERM STUDY OF THE SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: Extension Study Of Tanezumab In Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091016; P3 LONG TERM SAFETY EXTENSION (Other: Alias Study Number)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis
Keywords: Tanezumab OA arthritis
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tanezumab 10 mg (Experimental): Tanezumab 10 mg
  Interventions: Biological: tanezumab
- Tanezumab 5 mg (Experimental): Tanezumab 5 mg
  Interventions: Biological: tanezumab
- Tanezumab 2.5 mg (Experimental): Tanezumab 2.5 mg
  Interventions: Biological: tanezumab

INTERVENTIONS:
Biological: tanezumab — Tanezumab 10 mg
  Other Names: RN624
  Arms: Tanezumab 10 mg
Biological: tanezumab — Tanezumab 5 mg
  Other Names: RN624
  Arms: Tanezumab 5 mg
Biological: tanezumab — Tanezumab 2.5 mg
  Other Names: RN624
  Arms: Tanezumab 2.5 mg

SUMMARY:
Safety extension study of Phase 3 Osteoarthritis trials with Tanezumab

DETAILED DESCRIPTION:
This study was terminated on 27 October 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in previous (specific) Phase 3 trials of Tanezumab in osteoarthritis

Exclusion Criteria:

* Willing to comply with scheduled visits and treatment plan Is medically fit to participate in the trial in the judgement of the Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2147 (Actual)
Dates: Start 2009-02-06 (Actual); Primary Completion 2010-11-02 (Actual); Study Completion 2011-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (223):
- United States (223):
  - Pinncale Research Group, LLC, Anniston, Alabama
  - Anniston Medical Clinic, PC, Anniston, Alabama
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Greystone Medical Center, Birmingham, Alabama
  - Saadat Ansari, MD Office, Huntsville, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Clinical Research Advantage, Inc./Mesa Family Medical Center, PC, Mesa, Arizona
  - Clinical Research Advantage, Inc./Central Arizona Medical Associates, PC, Mesa, Arizona
  - Novara Clinical Research, Mesa, Arizona
  - Clinical Research Advantage, Inc., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Paradise Valley, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Clincial Research Advantage, Inc/Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research Advantage, Inc., Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Paradigm Clinical, Inc., Tucson, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Joseph's Mercy Clinic, Hot Springs, Arkansas
  - Osteoporosis Medical Center, Beverly Hills, California
  - Providence Clinical Research, Burbank, California
  - eStudySite, Chula Vista, California
  - Colorado Hematology - Oncology, Englewood, California
  - Colorado Orthopedic Consultants, PC, Englewood, California
  - Arthritis Medical Clinic of North County, Inc., Escondido, California
  - Edinger Medical Group Clinical Research, Fountain Valley, California
  - Valley Research, Fresno, California
  - Talbert Medical Group, Huntington Beach, California
  - Lakewood Orthopedic Medical & Surgical Group, Lakewood, California
  - High Desert Medical Group Research for Life, Lancaster, California
  - Premiere Clinical Research, LLC, Long Beach, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Del Carmen Medical Center, Reseda, California
  - Probe Clinical Research, Corp., Santa Ana, California
  - Trinity Clinical Trials, Santa Ana, California
  - Office of Lawrence P McAdam, MD, Thousand Oaks, California
  - Westlake Medical Research, Westlake Village, California
  - Colorado Orthopedic Consultants, PC, Aurora, Colorado
  - Peak Anesthesia and Pain Management, Centennial, Colorado
  - Denver Internal Medicine Group, Denver, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Advanced Orthopedic and Sports Medicine, Denver, Colorado
  - American Clinical Research, LLC, Englewood, Colorado
  - Orthopaedic Physicians Of Colorado, P.C., Englewood, Colorado
  - University Parks Hematology/Oncology, Englewood, Colorado
  - Advanced Orthopedic and Sports Medicine, Parker, Colorado
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Norwalk Medical Group, Norwalk, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - HeartCare (Private Practice), Bradenton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - In Vivo Clinical Research, Inc, Doral, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - Pharmax Research Clinic, Inc, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Compass Research, LLC, Orlando, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research Incorporated, Pembroke Pines, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Progressive Medical Research, Port Orange, Florida
  - HeartCare Research, Sarasota, Florida
  - Dale G. Bramlet, MD, P.L., St. Petersburg, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Jefrey D. Lieberman, MD, Decatur, Georgia
  - Early Family Practice Center, Fort Valley, Georgia
  - Northeast Georgia Diagnostic Clinic, LLC, Gainesville, Georgia
  - Marietta Rheumatology Associates, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Sonora Clinical Research, LLC., Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Illinois Bone and Joint Institute, LLC, Morton Grove, Illinois
  - The Arthritis Center, Springfield, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network, Fishers, Indiana
  - Memorial Medical Group Clinical Research Institute, South Bend, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Pasadena Pharmacy, Lexington, Kentucky
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Bluegrass Community Research, Inc, Lexington, Kentucky
  - David H. Neustadt, MD, Louisville, Kentucky
  - L-Marc Research Center, Louisville, Kentucky
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - The Baton Rouge Clinic, Baton Rouge, Louisiana
  - Stanocola Medical Center, Baton Rouge, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Arthritis Treatment Center, Frederick, Maryland
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Miray Medical Center, Brockton, Massachusetts
  - Mansfield Health Center, Mansfield, Massachusetts
  - Arthritis Associates Inc., Peabody, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Ann Arbor Clinical Research, Ann Arbor, Michigan
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - MAPS Applied Research Center Inc., Edina, Minnesota
  - Medical Advanced Pain Specialists, Edina, Minnesota
  - Planters Clinic, Port Gibson, Mississippi
  - St. John's Clinic - Neurology, Springfield, Missouri
  - St. John's Medical Research Institute, Inc., Springfield, Missouri
  - Medex Healthcare Research, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Midwest Minor Medical, Omaha, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Diagnostic Center of Medicine, Henderson, Nevada
  - Independent Clinical Researchers, Las Vegas, Nevada
  - Wolfson Medical Center, Las Vegas, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical, Las Vegas, Nevada
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - Office of Dr. Danka Michaels, MD, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Incorporated, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Medical Associates, Brooklyn, New York
  - Medex Healthcare Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Prem C. Chatpar, MD, LLC, Plainview, New York
  - AAIR Research Center, Rochester, New York
  - Office of Dr. Andrew Porges, Roslyn, New York
  - SPRI Bronx LLC, The Bronx, New York
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Carolina Bone & Joint, PA, Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Odyssey Research, Fargo, North Dakota
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - Consultants for Clinical Research Incorporated, Cincinnati, Ohio
  - Ohio GI and Liver Institute, Cincinnati, Ohio
  - Hilltop Medical Research Center, Cincinnati, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - PHP Center for Clinical Research, Dayton, Ohio
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Orthopaedic & Sports Medicine Consultants, Middletown, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Pharmacotherapy Research Associates,Inc, Zanesville, Ohio
  - Physicians' Research, Inc, Zanesville, Ohio
  - Primecare of Southeastern Ohio, Inc, Zanesville, Ohio
  - Cor Clinical Research, LLC, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - The Family Healthcare Center, PA, Clinton, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - The Carolina Center for Rheumatology and Arthritis Care, PA, Rock Hill, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - State of Franklin Healthcare Associates, PLLC, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Capitol Medical Clinic, Austin, Texas
  - Walter F. Chase, MD, PA, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - North Texas Joint Care, PA, Dallas, Texas
  - Crown Imaging, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Radiant Research, Dallas, Texas
  - O. David Taunton, Jr, MD, Grapevine, Texas
  - Asif Cochinwala, MD, PA, Houston, Texas
  - Foundation for Southwest Orthopedic Research, Houston, Texas
  - One Step Diagnostic, Houston, Texas
  - Southwest Orthopedic Group, Houston, Texas
  - The Neurology Center, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Gill Orthopedic Center, Lubbock, Texas
  - Robert R. King, M.D., Lubbock, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Texas Arthritis Research Center, PA, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Spring Family Practice Associates PA, Spring, Texas
  - AZ Clinical Research, Sugar Land, Texas
  - Spring Clinical Research, Sugar Land, Texas
  - Sugar Land Med-Ped, P.A., Sugar Land, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Aspen Clinical Research, Orem, Utah
  - Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Incorporated/Foothill Family Clinic South, Salt Lake City, Utah
  - Commonwealth Orthopaedics and Rehabilitation, PC, Arlington, Virginia
  - IntegraTrials, LLC, Arlington, Virginia
  - Virginia Hospital Center, Arlington, Virginia
  - Charlottesville Medical Research, Charlottesville, Virginia
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Office of Doris M. Rice, MD, FACR, Portsmouth, Virginia
  - HhypotheTest, LLC, Roanoke, Virginia
  - Empirical Clinical Trials, Selah, Washington
  - Arthritis Northwest, Spokane, Washington
  - Clinical Trials Northwest, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091016&StudyName=Extension%20Study%20Of%20Tanezumab%20In%20Osteoarthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants randomized and treated with study medication in parent studies A4091011 (NCT00733902), A4091014 (NCT00744471), A4091015 (NCT00830063) and A4091018 (NCT00863304) who had completed the treatment period or discontinued due to lack of efficacy were eligible to enroll in this study.
Pre-assignment Details: 533 participants who received placebo and 294 participants who received naproxen in parent studies were randomized to receive tanezumab 2.5, 5 or 10 milligram (mg) on Day 1. The remaining participants who received tanezumab in parent studies remained on the same dose they received in parent studies.
Groups:
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg intravenous infusion administered every 8 weeks for up to 64 weeks.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg intravenous infusion administered every 8 weeks for up to 64 weeks.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion administered every 8 weeks for up to 64 weeks.
Period: Overall Study
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Started | 525 | 832 | 790
Treated | 522 | 832 | 788
Completed | 0 | 0 | 0
Not Completed | 525 | 832 | 790
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 34 | 52 | 71
Not completed — Lack of Efficacy | 39 | 52 | 63
Not completed — Lost to Follow-up | 0 | 3 | 4
Not completed — Withdrawal by Subject | 47 | 72 | 64
Not completed — Protocol Violation | 2 | 6 | 5
Not completed — Randomized, but not treated | 3 | 0 | 2
Not completed — Study Terminated by Sponsor | 378 | 626 | 565
Not completed — Other | 21 | 21 | 16

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all participants who received at least 1 dose of intravenous study medication during this study, A4091016 (NCT00809783).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg | Total
Number analyzed (Participants) | 522 | 832 | 788 | 2142
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 29 | 43 | 32 | 104
  45 to 64 years | 298 | 466 | 455 | 1219
  Greater than or equal to 65 years | 195 | 323 | 301 | 819
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 522 | 474 | 1304
  Male | 214 | 310 | 314 | 838

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: AE:any untoward medical occurrence in participant who received study medication without regard to possibility of causal relationship. SAE:an AE resulting in any of following outcomes or deemed significant for any other reason:death;initial or prolonged inpatient hospitalization;life-threatening experience(immediate risk of dying);persistent or significant disability/incapacity;congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 112 days after last dose that were absent before treatment in this study or that worsened relative to pretreatment state. AEs included both SAEs and all non-SAEs.
Time Frame: A4091016: Baseline (Day 1) up to 112 days after last dose of study medication (up to Week 80)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
Participants
  AEs | 363 | 573 | 547
  SAEs | 47 | 73 | 96

2. Primary Outcome: Number of Participants With Abnormal Laboratory Findings
Description: Hemoglobin(Hgb),hematocrit,red blood cell(RBC):less than(<)0.8*lower limit of normal(LLN),MCV,MCH,MCHC<0.9*LLN or >1.1*ULN,platelet:<0.5*LLN or >1.75*upper limit of normal(ULN),white blood cell(WBC):<0.6*LLN or >1.5*ULN,lymphocyte,neutrophil,total neutrophil:<0.8*LLN or>1.2*ULN,basophil,eosinophil,monocyte:>1.2*ULN;total,direct bilirubin>1.5*ULN,aspartate aminotransferase,alanine aminotransferase,gamma-glutamyl transferase,LDH,alkaline phosphatase:> 3.0*ULN,total protein,albumin:<0.8*LLN or >1.2*ULN;blood urea nitrogen,creatinine:>1.3*ULN,uric acid>1.2*ULN;cholesterol,triglycerides>1.3*ULN;sodium <0.95*LLN or >1.05*ULN,potassium,chloride,calcium,magnesium,bicarbonate:<0.9*LLN or >1.1*ULN,phosphate<0.8*LLN or>1.2*ULN;glucose <0.6*LLN or >1.5*ULN,glycosylated Hgb >1.3*ULN,creatine kinase>2.0*ULN;urine(specific gravity <1.003or>1.030,pH <4.5or>8,glucose,ketone,protein,blood/Hgb,bilirubin,leukocyte esterase,crystals>=1,RBC,WBC >1.5*ULN,epithelial cell>=6,casts,hyaline cast>1,bacteria>20).
Time Frame: A4091016: Day 1 up to Week 80
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study, A4091016 (NCT00809783). "Overall number of participants analyzed" signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 516 | 810 | 767
Participants | 439 | 679 | 624

3. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: Following parameters were analyzed for ECG abnormality: PR interval, QRS interval, QT interval, QT interval corrected using the Fridericia's formula (QTcF), QT interval corrected using the Bazett's formula (QTcB), RR interval and VR interval. Number of participants with clinically significant abnormal ECG findings were judged by investigator and reported as adverse events were presented.
Time Frame: A4091016: Baseline (Day 1) up to Week 80
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study, A4091016 (NCT00809783).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
Participants | 14 | 33 | 17

4. Secondary Outcome: Change From Parent Study Baseline in Neuropathy Impairment Score (NIS) at Week 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: NIS constitutes sum of 37 standard items of neuromuscular examination used to assess muscle strength, reflexes and sensation. Each item is scored separately for left and right sides. Components of muscle weakness (24 items) scored on a scale: 0 (normal) to 4 (paralysis), with higher score=more weakness; components of reflexes and sensation (13 items) scored on a scale: 0= normal, 1= decreased or 2= absent. Total NIS score range 0 (no impairment) to 244 (maximum impairment), higher score = more impairment. Parent study baseline value calculated as average of pre-dose measurements of participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: Baseline of the parent study (A4091011, A4091014, A4091015, A4091018); A4091016: Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: ITT population. Last observation carried forward (LOCF) method was used to impute missing values. "Overall number of participants analyzed" signifies those participants who were evaluable for this measure. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 785
units on a scale
  Parent Study Baseline | 1.06 (3.16) | 0.95 (2.55) | 1.09 (3.08)
  Change at Week 4: number analyzed (Participants) | 502 | 792 | 756
  Change at Week 4 | -0.10 (0.97) | -0.04 (1.15) | -0.12 (1.91)
  Change at Week 8: number analyzed (Participants) | 515 | 818 | 771
  Change at Week 8 | -0.04 (1.60) | -0.02 (1.43) | -0.03 (1.72)
  Change at Week 16: number analyzed (Participants) | 515 | 819 | 772
  Change at Week 16 | -0.07 (1.51) | -0.03 (1.79) | -0.07 (2.00)
  Change at Week 24: number analyzed (Participants) | 516 | 819 | 773
  Change at Week 24 | -0.09 (1.65) | -0.04 (1.74) | -0.12 (1.82)
  Change at Week 32: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 32 | -0.05 (1.44) | -0.02 (1.66) | -0.05 (1.79)
  Change at Week 40: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 40 | -0.01 (2.57) | 0.02 (1.62) | -0.11 (1.93)
  Change at Week 48: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 48 | -0.04 (2.47) | -0.03 (1.54) | -0.11 (1.89)
  Change at Week 56: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 56 | -0.02 (2.61) | -0.04 (1.56) | -0.11 (1.89)
  Change at Week 64: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 64 | -0.04 (2.58) | -0.07 (1.59) | -0.12 (1.89)
  Change at Week 72: number analyzed (Participants) | 518 | 821 | 774
  Change at Week 72 | -0.04 (2.57) | -0.05 (1.59) | -0.11 (1.87)

5. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) for Tanezumab
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). Same participant may have positive ADA result at more than 1 time point.
Time Frame: A4091016: Day 1, Week 16, 24, 40, 56, 72, 80 or Early Termination (ET: anytime till Week 80)
Population: ITT population. "Overall number of participants analyzed" signifies those participants who were evaluable for this measure at any time point. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 492 | 775 | 733
Participants
  Day 1: number analyzed (Participants) | 88 | 114 | 117
  Day 1 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 421 | 675 | 636
  Week 16 | 1 | 1 | 4
  Week 24: number analyzed (Participants) | 351 | 531 | 472
  Week 24 | 0 | 1 | 3
  Week 40: number analyzed (Participants) | 197 | 237 | 200
  Week 40 | 1 | 0 | 0
  Week 56: number analyzed (Participants) | 59 | 63 | 45
  Week 56 | 2 | 0 | 1
  Week 72: number analyzed (Participants) | 3 | 5 | 1
  Week 72 | 0 | 0 | 0
  Week 80 or ET: number analyzed (Participants) | 402 | 641 | 605
  Week 80 or ET | 2 | 2 | 5

6. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline to Week 80 in Physical Examination Findings
Description: Physical examination included examination of following sites in addition to general examination: abdomen, ears, extremities, eyes, head, heart, musculoskeletal, neck, nose, skin, throat and thyroid. Clinically significant changes were judged by investigator.
Time Frame: Baseline (Day 1) up to Week 80
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
Participants | 26 | 48 | 53

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Vital Signs
Description: Following parameters were analyzed for examination of vital signs: body temperature, blood pressure, heart rate and respiratory rate. Number of participants with clinically significant abnormality in vital signs were judged by investigator and reported as adverse events were presented.
Time Frame: A4091016: Baseline (Day 1) up to Week 80
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
participants | 12 | 13 | 23

8. Secondary Outcome: Change From Parent Study Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or hip joint during past 48 hours. The WOMAC pain score is calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (minimum pain) to 10 (maximum pain), where higher scores indicate higher pain. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: Baseline of the parent study (A4091011, A4091014, A4091015, A4091018); A4091016: Week 4, 8, 16, 24, 32, 40, 48,56, 64, 72, 80, 88, 96, 104
Population: ITT population. LOCF method was used to impute missing values. "Overall number of participants analyzed" signifies those participants who were evaluable for this measure. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 80, 88, 96 and 104 were not reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
units on a scale
  Parent Study Baseline | 7.20 (1.43) | 7.20 (1.40) | 7.19 (1.47)
  Change at Week 4 | -4.47 (2.31) | -4.47 (2.41) | -4.52 (2.48)
  Change at Week 8 | -4.04 (2.52) | -4.19 (2.44) | -4.45 (2.53)
  Change at Week 16 | -3.98 (2.49) | -4.08 (2.47) | -4.29 (2.57)
  Change at Week 24 | -3.88 (2.52) | -4.03 (2.49) | -4.17 (2.62)
  Change at Week 32 | -3.76 (2.56) | -3.95 (2.56) | -4.10 (2.64)
  Change at Week 40 | -3.73 (2.59) | -3.90 (2.56) | -4.07 (2.66)
  Change at Week 48 | -3.71 (2.60) | -3.87 (2.55) | -4.05 (2.66)
  Change at Week 56 | -3.72 (2.59) | -3.87 (2.55) | -4.03 (2.67)
  Change at Week 64 | -3.71 (2.60) | -3.86 (2.56) | -4.02 (2.67)
  Change at Week 72 | -3.71 (2.60) | -3.87 (2.55) | -4.02 (2.67)

9. Secondary Outcome: Change From Parent Study Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index knee or hip joint during past 48 hours. The WOMAC physical function score is calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicate worse function. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 518 | 830 | 784
units on a scale
  Parent Study Baseline | 6.75 (1.62) | 6.81 (1.57) | 6.81 (1.61)
  Change at Week 4 | -3.93 (2.39) | -4.05 (2.38) | -4.10 (2.44)
  Change at Week 8 | -3.47 (2.59) | -3.75 (2.45) | -4.05 (2.49)
  Change at Week 16 | -3.45 (2.57) | -3.65 (2.46) | -3.87 (2.55)
  Change at Week 24 | -3.34 (2.60) | -3.60 (2.50) | -3.74 (2.60)
  Change at Week 32 | -3.21 (2.65) | -3.51 (2.54) | -3.67 (2.62)
  Change at Week 40 | -3.18 (2.66) | -3.45 (2.53) | -3.64 (2.65)
  Change at Week 48 | -3.15 (2.66) | -3.44 (2.52) | -3.61 (2.65)
  Change at Week 56 | -3.16 (2.65) | -3.43 (2.53) | -3.59 (2.65)
  Change at Week 64 | -3.16 (2.65) | -3.42 (2.53) | -3.59 (2.65)
  Change at Week 72 | -3.16 (2.66) | -3.42 (2.53) | -3.59 (2.65)

10. Secondary Outcome: Change From Parent Study Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee/hip affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good and 5 = very poor. Higher scores indicate worse condition. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: ITT population. LOCF method was used to impute missing values. '"Overall number of participants analyzed" = participants who were evaluable for this measure. "Number Analyzed" = participants who were evaluable for this measure at given time points for each group, respectively. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 80, 88, 96, 104 were not reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 829 | 785
units on a scale
  Parent Study Baseline | 3.45 (0.58) | 3.43 (0.60) | 3.45 (0.60)
  Change at Week 4: number analyzed (Participants) | 519 | 828 | 785
  Change at Week 4 | -1.18 (0.93) | -1.22 (0.97) | -1.22 (0.99)
  Change at Week 8 | -0.98 (0.99) | -1.08 (0.96) | -1.17 (1.00)
  Change at Week 16 | -0.94 (0.95) | -1.06 (0.98) | -1.10 (0.99)
  Change at Week 24 | -0.88 (0.93) | -1.01 (0.99) | -1.03 (1.05)
  Change at Week 32 | -0.88 (0.95) | -1.00 (1.00) | -1.01 (1.06)
  Change at Week 40 | -0.85 (0.98) | -0.94 (1.00) | -0.97 (1.07)
  Change at Week 48 | -0.83 (0.98) | -0.94 (1.01) | -0.97 (1.08)
  Change at Week 56 | -0.84 (0.97) | -0.94 (1.01) | -0.96 (1.08)
  Change at Week 64 | -0.83 (0.97) | -0.93 (1.01) | -0.96 (1.09)
  Change at Week 72 | -0.83 (0.97) | -0.93 (1.01) | -0.96 (1.09)

11. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: OMERACT-OARSI response:>=50 percent(%) improvement from parent study baseline and absolute change from parent study baseline of >=2 units at given week in WOMAC pain or physical function subscale or >=20% improvement from parent study baseline and absolute change from parent study baseline of >=1 unit at given week in at least 2 of following 3 items: 1)WOMAC pain subscale, 2)WOMAC physical function subscale, 3)PGA of osteoarthritis (score: 1-5, higher score=more affected).WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score:0-10, higher score=higher pain/difficulty).
Time Frame: A4091016: Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study, A4091016 (NCT00809783). LOCF method was used to impute missing values. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 80, 88, 96 and 104 were not reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
percentage of participants
  Week 4 | 86.8 [83.9 to 89.7] | 88.5 [86.3 to 90.6] | 86.0 [83.6 to 88.5]
  Week 8 | 80.3 [76.9 to 83.7] | 83.5 [81.0 to 86.1] | 85.0 [82.5 to 87.5]
  Week 16 | 80.1 [76.7 to 83.5] | 83.2 [80.6 to 85.7] | 82.9 [80.2 to 85.5]
  Week 24 | 77.4 [73.8 to 81.0] | 82.0 [79.4 to 84.6] | 81.5 [78.8 to 84.2]
  Week 32 | 75.1 [71.4 to 78.8] | 79.9 [77.2 to 82.6] | 80.2 [77.4 to 83.0]
  Week 40 | 75.1 [71.4 to 78.8] | 79.3 [76.6 to 82.1] | 79.9 [77.2 to 82.7]
  Week 48 | 74.5 [70.8 to 78.3] | 79.4 [76.7 to 82.2] | 79.6 [76.8 to 82.4]
  Week 56 | 74.9 [71.2 to 78.6] | 79.3 [76.6 to 82.1] | 79.2 [76.4 to 82.0]
  Week 64 | 74.5 [70.8 to 78.3] | 79.2 [76.4 to 82.0] | 79.2 [76.4 to 82.0]
  Week 72 | 74.5 [70.8 to 78.3] | 79.2 [76.4 to 82.0] | 79.2 [76.4 to 82.0]

12. Secondary Outcome: Percentage of Participants With at Least 30%, 50%, 70% and 90% Reduction From Parent Study Baseline in WOMAC Pain Subscale Score
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
percentage of participants
  Week 4: >=30% reduction | 83.6 | 82.6 | 81.3
  Week 4: >=50% reduction | 70.1 | 68.7 | 69.9
  Week 4: >=70% reduction | 48.2 | 50.9 | 48.9
  Week 4: >=90% reduction | 21.6 | 23.1 | 24.2
  Week 8: >=30% reduction | 75.5 | 78.6 | 81.4
  Week 8: >=50% reduction | 64.0 | 63.9 | 68.3
  Week 8: >=70% reduction | 41.6 | 43.2 | 48.2
  Week 8: >=90% reduction | 18.9 | 20.7 | 25.4
  Week 16: >=30% reduction | 76.5 | 76.9 | 79.7
  Week 16: >=50% reduction | 63.0 | 61.4 | 66.5
  Week 16: >=70% reduction | 39.1 | 42.0 | 45.7
  Week 16: >=90% reduction | 18.1 | 18.8 | 21.8
  Week 24: >=30% reduction | 73.6 | 77.4 | 77.1
  Week 24: >=50% reduction | 60.3 | 61.6 | 63.3
  Week 24: >=70% reduction | 38.3 | 40.3 | 45.5
  Week 24: >=90% reduction | 16.8 | 19.3 | 21.5
  Week 32: >=30% reduction | 72.6 | 75.5 | 75.9
  Week 32: >=50% reduction | 57.4 | 59.8 | 62.7
  Week 32: >=70% reduction | 36.8 | 42.2 | 43.8
  Week 32: >=90% reduction | 16.6 | 19.1 | 20.4
  Week 40: >=30% reduction | 71.5 | 74.4 | 75.9
  Week 40: >=50% reduction | 57.0 | 58.1 | 61.7
  Week 40: >=70% reduction | 37.0 | 41.2 | 43.8
  Week 40: >=90% reduction | 15.8 | 19.4 | 19.7
  Week 48: >=30% reduction | 71.1 | 73.9 | 75.4
  Week 48: >=50% reduction | 56.6 | 58.5 | 61.4
  Week 48: >=70% reduction | 35.8 | 40.0 | 43.4
  Week 48: >=90% reduction | 15.4 | 18.3 | 19.5
  Week 56: >=30% reduction | 71.5 | 73.8 | 75.2
  Week 56: >=50% reduction | 57.0 | 58.1 | 61.1
  Week 56: >=70% reduction | 36.0 | 39.8 | 43.2
  Week 56: >=90% reduction | 15.6 | 19.0 | 19.2
  Week 64: >=30% reduction | 71.3 | 73.8 | 75.2
  Week 64: >=50% reduction | 56.8 | 58.2 | 61.1
  Week 64: >=70% reduction | 36.2 | 39.8 | 43.2
  Week 64: >=90% reduction | 15.6 | 19.0 | 19.2
  Week 72: >=30% reduction | 71.3 | 73.8 | 75.2
  Week 72: >=50% reduction | 56.8 | 58.2 | 61.0
  Week 72: >=70% reduction | 36.2 | 39.8 | 43.1
  Week 72: >=90% reduction | 15.6 | 19.0 | 19.2

13. Secondary Outcome: Number of Participants With Cumulative Reduction From Parent Study Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16, 24, 56 and 104
Description: as for outcome 8
Time Frame: Baseline of the parent study (A4091011, A4091014, A4091015, A4091018); A4091016: Week 16, 24, 56, 104
Population: ITT population. LOCF method was used to impute missing values. "Overall number of participants analyzed" signifies those participants who were evaluable for this measure. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 104 were not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
Participants
  Week 16: Greater than 0% reduction | 478 | 782 | 733
  Week 16: >=10% reduction | 462 | 750 | 708
  Week 16: >=20% reduction | 431 | 701 | 665
  Week 16: >=30% reduction | 397 | 639 | 626
  Week 16: >=40% reduction | 358 | 573 | 577
  Week 16: >=50% reduction | 327 | 510 | 522
  Week 16: >=60% reduction | 267 | 432 | 453
  Week 16: >=70% reduction | 203 | 349 | 359
  Week 16: >=80% reduction | 149 | 264 | 271
  Week 16: >=90 reduction | 94 | 156 | 171
  Week 16: 100% reduction | 30 | 68 | 78
  Week 24: Greater than 0% reduction | 477 | 782 | 734
  Week 24: >=10% reduction | 457 | 750 | 703
  Week 24: >=20% reduction | 419 | 692 | 655
  Week 24: >=30% reduction | 382 | 643 | 605
  Week 24: >=40% reduction | 352 | 567 | 552
  Week 24: >=50% reduction | 313 | 512 | 497
  Week 24: >=60% reduction | 264 | 425 | 432
  Week 24: >=70% reduction | 199 | 335 | 357
  Week 24: >=80% reduction | 141 | 255 | 271
  Week 24: >=90% reduction | 87 | 160 | 169
  Week 24: 100% reduction | 29 | 69 | 66
  Week 56: Greater than 0% reduction | 470 | 773 | 726
  Week 56: >=10% reduction | 449 | 735 | 689
  Week 56: >=20% reduction | 409 | 677 | 640
  Week 56: >=30% reduction | 371 | 613 | 590
  Week 56: >=40% reduction | 334 | 545 | 538
  Week 56: >=50% reduction | 296 | 483 | 480
  Week 56: >=60% reduction | 249 | 404 | 414
  Week 56: >=70% reduction | 187 | 331 | 339
  Week 56: >=80% reduction | 128 | 250 | 255
  Week 56: >=90% reduction | 81 | 158 | 151
  Week 56: 100% reduction | 30 | 63 | 69

14. Secondary Outcome: Percentage of Participants With Improvement of at Least 2 Points From Parent Study Baseline in Patient Global Assessment (PGA) of Osteoarthritis
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee/hip affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good and 5 = very poor. Higher scores indicated worse pain. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 829 | 785
percentage of participants
  Week 4: number analyzed (Participants) | 519 | 828 | 785
  Week 4 | 37.6 [33.4 to 41.7] | 36.6 [33.3 to 39.9] | 37.3 [33.9 to 40.7]
  Week 8 | 28.9 [25.0 to 32.8] | 31.0 [27.9 to 34.1] | 34.9 [31.6 to 38.2]
  Week 16 | 29.9 [25.9 to 33.8] | 30.8 [27.6 to 33.9] | 31.7 [28.5 to 35.0]
  Week 24 | 25.8 [22.1 to 29.6] | 28.7 [25.6 to 31.8] | 32.4 [29.1 to 35.6]
  Week 32 | 25.8 [22.1 to 29.6] | 28.3 [25.3 to 31.4] | 31.0 [27.7 to 34.2]
  Week 40 | 25.4 [21.7 to 29.2] | 26.1 [23.1 to 29.0] | 29.9 [26.7 to 33.1]
  Week 48 | 24.7 [21.0 to 28.4] | 26.7 [23.6 to 29.7] | 30.3 [27.1 to 33.5]
  Week 56 | 24.7 [21.0 to 28.4] | 26.5 [23.5 to 29.5] | 30.2 [27.0 to 33.4]
  Week 64 | 24.7 [21.0 to 28.4] | 26.3 [23.3 to 29.3] | 30.1 [26.9 to 33.3]
  Week 72 | 24.7 [21.0 to 28.4] | 26.3 [23.3 to 29.3] | 30.1 [26.9 to 33.3]

15. Secondary Outcome: Change From Parent Study Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: WOMAC stiffness subscale: questionnaire used to assess amount of stiffness experienced due to osteoarthritis in index joint during past 48 hours. The WOMAC stiffness score is calculated as mean of scores from 2 individual questions scored on NRS of 0 (minimum stiffness) to 10 (maximum stiffness), higher scores indicate higher stiffness. Total score range for WOMAC stiffness subscale score =0 (minimum stiffness) to 10 (maximum stiffness), higher scores indicate higher stiffness. Stiffness is defined as sensation of decreased ease in movement of knee/hip. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: ITT population. LOCF method was used to impute missing values. '"Overall number of participants analyzed" = participants who were evaluable for this measure. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 80, 88, 96, 104 were not reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
units on a scale
  Parent Study Baseline | 7.00 (1.83) | 7.06 (1.78) | 7.05 (1.85)
  Change at Week 4 | -4.14 (2.66) | -4.29 (2.63) | -4.36 (2.73)
  Change at Week 8 | -3.69 (2.81) | -4.00 (2.71) | -4.33 (2.76)
  Change at Week 16 | -3.56 (2.83) | -3.85 (2.70) | -4.10 (2.84)
  Change at Week 24 | -3.46 (2.78) | -3.81 (2.71) | -4.02 (2.91)
  Change at Week 32 | -3.35 (2.83) | -3.73 (2.76) | -3.91 (2.95)
  Change at Week 40 | -3.29 (2.86) | -3.65 (2.79) | -3.90 (2.95)
  Change at Week 48 | -3.25 (2.87) | -3.64 (2.77) | -3.87 (2.96)
  Change at Week 56 | -3.27 (2.85) | -3.63 (2.77) | -3.85 (2.96)
  Change at Week 64 | -3.26 (2.86) | -3.63 (2.77) | -3.85 (2.96)
  Change at Week 72 | -3.26 (2.86) | -3.63 (2.77) | -3.85 (2.96)

16. Secondary Outcome: Change From Parent Study Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee or hip. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 (minimum difficulty) to 10 (maximum difficulty), where higher score indicates worse response. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
units on a scale
  Parent Study Baseline | 6.98 (1.44) | 7.02 (1.43) | 7.01 (1.46)
  Change at Week 4 | -4.18 (2.31) | -4.27 (2.33) | -4.33 (2.41)
  Change at Week 8 | -3.74 (2.49) | -3.98 (2.39) | -4.28 (2.45)
  Change at Week 16 | -3.67 (2.49) | -3.86 (2.40) | -4.09 (2.51)
  Change at Week 24 | -3.57 (2.50) | -3.81 (2.42) | -3.98 (2.57)
  Change at Week 32 | -3.45 (2.55) | -3.73 (2.48) | -3.89 (2.60)
  Change at Week 40 | -3.41 (2.57) | -3.67 (2.49) | -3.87 (2.61)
  Change at Week 48 | -3.38 (2.58) | -3.65 (2.47) | -3.85 (2.62)
  Change at Week 56 | -3.39 (2.57) | -3.64 (2.47) | -3.83 (2.62)
  Change at Week 64 | -3.39 (2.58) | -3.64 (2.48) | -3.82 (2.63)
  Change at Week 72 | -3.38 (2.58) | -3.64 (2.48) | -3.82 (2.62)

17. Secondary Outcome: Change From Parent Study Baseline For Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Downstairs at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: Participants answered: "How much pain have you had going up or down the stairs?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicates more pain. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 518 | 830 | 785
units on a scale
  Parent Study Baseline | 8.14 (1.48) | 8.11 (1.48) | 8.16 (1.51)
  Change at Week 4: number analyzed (Participants) | 518 | 830 | 784
  Change at Week 4 | -4.60 (2.61) | -4.54 (2.74) | -4.73 (2.74)
  Change at Week 8 | -4.15 (2.83) | -4.25 (2.75) | -4.69 (2.83)
  Change at Week 16 | -4.01 (2.79) | -4.05 (2.85) | -4.46 (2.84)
  Change at Week 24 | -3.85 (2.86) | -3.97 (2.86) | -4.33 (2.91)
  Change at Week 32 | -3.76 (2.87) | -3.87 (2.91) | -4.24 (2.92)
  Change at Week 40 | -3.70 (2.92) | -3.81 (2.93) | -4.21 (2.94)
  Change at Week 48 | -3.72 (2.88) | -3.78 (2.93) | -4.19 (2.95)
  Change at Week 56 | -3.74 (2.86) | -3.80 (2.94) | -4.16 (2.94)
  Change at Week 64 | -3.75 (2.87) | -3.79 (2.94) | -4.16 (2.94)
  Change at Week 72 | -3.74 (2.87) | -3.79 (2.94) | -4.15 (2.95)

18. Secondary Outcome: Change From Parent Study Baseline For Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96 and 104
Description: Participants answered: "How much pain have you had when walking on a flat surface?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicates more pain. Parent study baseline value calculated as average of pre-dose measurements of the participants from study A4091011, A4091014, A4091015 and A4091018.
Time Frame: as for outcome 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 519 | 831 | 785
units on a scale
  Parent Study Baseline | 7.22 (1.67) | 7.10 (1.63) | 7.10 (1.66)
  Change at Week 4 | -4.51 (2.54) | -4.36 (2.59) | -4.38 (2.67)
  Change at Week 8 | -4.07 (2.78) | -4.03 (2.65) | -4.24 (2.73)
  Change at Week 16 | -3.96 (2.74) | -3.85 (2.74) | -4.12 (2.84)
  Change at Week 24 | -3.88 (2.79) | -3.83 (2.72) | -3.97 (2.85)
  Change at Week 32 | -3.74 (2.78) | -3.77 (2.78) | -3.88 (2.87)
  Change at Week 40 | -3.70 (2.83) | -3.68 (2.80) | -3.86 (2.89)
  Change at Week 48 | -3.72 (2.82) | -3.65 (2.78) | -3.83 (2.90)
  Change at Week 56 | -3.71 (2.81) | -3.66 (2.78) | -3.81 (2.91)
  Change at Week 64 | -3.72 (2.82) | -3.65 (2.79) | -3.80 (2.91)
  Change at Week 72 | -3.71 (2.82) | -3.65 (2.79) | -3.80 (2.91)

19. Secondary Outcome: Percentage of Participants Who Used Concomitant Analgesic Medication
Description: United States Food and Drug Administration (FDA) approved analgesics (over-the-counter or prescription) were permitted as concomitant medications to relieve the pain of osteoarthritis. These medications included opioids, topical analgesics, non-steroidal anti inflammatory drugs (NSAIDs), capsaicin products, oral/injectable corticosteroids and viscosupplementation (hyaluronan) and were prescribed as per investigator's discretion.
Time Frame: Week 1-4, 5-8, 9-16, 17-24, 25-32, 33-40, 41-48, 49-56, 57-64, 65-72, 73-80, 81-88, 89-96, 97-104, 105-112
Population: ITT population. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively. Efficacy results were not collected beyond Week 72 due to clinical hold. Therefore, results for Week 73-80, 81-88, 89-96, 97-104 and 105-112 were not reported.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
percentage of participants
  Week 1-4 | 31.8 | 28.7 | 31.1
  Week 5-8: number analyzed (Participants) | 518 | 817 | 773
  Week 5-8 | 33.2 | 35.4 | 32.1
  Week 9-16: number analyzed (Participants) | 509 | 792 | 760
  Week 9-16 | 39.5 | 44.4 | 45.3
  Week 17-24: number analyzed (Participants) | 480 | 744 | 708
  Week 17-24 | 40.4 | 43.4 | 47.5
  Week 25-32: number analyzed (Participants) | 415 | 634 | 589
  Week 25-32 | 40.7 | 34.1 | 30.9
  Week 33-40: number analyzed (Participants) | 331 | 469 | 433
  Week 33-40 | 36.0 | 26.4 | 35.3
  Week 41-48: number analyzed (Participants) | 246 | 329 | 294
  Week 41-48 | 42.3 | 19.1 | 34.7
  Week 49-56: number analyzed (Participants) | 172 | 200 | 162
  Week 49-56 | 37.2 | 34.0 | 16.0
  Week 57-64: number analyzed (Participants) | 91 | 114 | 79
  Week 57-64 | 11.0 | 28.1 | 31.6
  Week 65-72: number analyzed (Participants) | 39 | 43 | 36
  Week 65-72 | 10.3 | 4.7 | 16.7

20. Secondary Outcome: Days Per Week of Concomitant Analgesic Medication Usage
Description: FDA approved analgesics (over-the-counter or prescription) were permitted as concomitant medications to relieve the pain of osteoarthritis. These medications included opioids, topical analgesics, NSAIDs, capsaicin products, oral/injectable corticosteroids and viscosupplementation (hyaluronan) and were prescribed at the discretion of the investigator.
Time Frame: Week 1-4, 5-8, 9-16, 17-24, 25-32, 33-40, 41-48, 49-56, 57-64, 65-72, 73-80, 81-88, 89-96, 97-104, 105-112
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
days per week
  Week 1-4 | 1.8 (2.98) | 1.6 (2.83) | 1.7 (2.85)
  Week 5-8: number analyzed (Participants) | 518 | 817 | 773
  Week 5-8 | 2.0 (3.13) | 1.9 (3.06) | 1.9 (3.05)
  Week 9-16: number analyzed (Participants) | 509 | 792 | 760
  Week 9-16 | 2.1 (3.09) | 2.0 (3.07) | 1.9 (3.00)
  Week 17-24: number analyzed (Participants) | 480 | 744 | 708
  Week 17-24 | 1.8 (2.93) | 1.7 (2.84) | 1.6 (2.74)
  Week 25-32: number analyzed (Participants) | 415 | 634 | 589
  Week 25-32 | 1.7 (2.89) | 1.4 (2.64) | 1.3 (2.58)
  Week 33-40: number analyzed (Participants) | 331 | 469 | 433
  Week 33-40 | 1.6 (2.80) | 1.1 (2.33) | 1.0 (2.31)
  Week 41-48: number analyzed (Participants) | 246 | 329 | 294
  Week 41-48 | 1.3 (2.59) | 0.8 (2.08) | 0.7 (1.94)
  Week 49-56: number analyzed (Participants) | 172 | 200 | 162
  Week 49-56 | 0.9 (2.03) | 0.8 (2.05) | 0.5 (1.59)
  Week 57-64: number analyzed (Participants) | 91 | 114 | 79
  Week 57-64 | 0.5 (1.66) | 0.4 (1.39) | 0.2 (0.67)
  Week 65-72: number analyzed (Participants) | 39 | 43 | 36
  Week 65-72 | 0.3 (0.97) | 0.0 (0.19) | 0.2 (1.13)

21. Other Pre Specified Outcome: Number of Participants Classified According to Number of Intravenous Doses of Study Medication
Description: Number of participants were reported based on the maximum number of intravenous doses of either tanezumab or placebo received.
Time Frame: A4091016: Baseline (Day 1) up to Week 64
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 522 | 832 | 788
Participants
  1 dose | 39 | 81 | 69
  2 doses | 91 | 161 | 164
  3 doses | 92 | 172 | 177
  4 doses | 78 | 158 | 141
  5 doses | 81 | 104 | 121
  6 doses | 76 | 79 | 62
  7 doses | 49 | 59 | 41
  8 doses | 13 | 13 | 11
  9 doses | 3 | 5 | 2

ADVERSE EVENTS:
Description: Participants may have experienced both non serious and SAE during study. Cases of osteonecrosis (ON) reported in this and other studies of this program, conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492.
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Serious Adverse Events (participants affected / at risk) | 47/522 | 73/832 | 96/788
Other Adverse Events (participants affected / at risk) | 280/522 | 412/832 | 408/788
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=522) | Tanezumab 5 mg (N=832) | Tanezumab 10 mg (N=788)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 3 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular failure (Cardiac disorders) | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 3
Oedema (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Chondrolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 22 | 25
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6 | 9 | 13
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=522) | Tanezumab 5 mg (N=832) | Tanezumab 10 mg (N=788)
Diarrhoea (Gastrointestinal disorders) | 7 | 18 | 8
Oedema peripheral (General disorders) | 22 | 52 | 57
Bronchitis (Infections and infestations) | 8 | 9 | 16
Nasopharyngitis (Infections and infestations) | 14 | 19 | 18
Sinusitis (Infections and infestations) | 15 | 26 | 21
Upper respiratory tract infection (Infections and infestations) | 36 | 42 | 29
Urinary tract infection (Infections and infestations) | 29 | 57 | 42
Contusion (Injury, poisoning and procedural complications) | 12 | 10 | 17
Fall (Injury, poisoning and procedural complications) | 26 | 23 | 40
Muscle strain (Injury, poisoning and procedural complications) | 12 | 12 | 19
Blood creatine phosphokinase increased (Investigations) | 15 | 14 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 | 116 | 121
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 22 | 37
Joint effusion (Musculoskeletal and connective tissue disorders) | 8 | 18 | 18
Joint swelling (Musculoskeletal and connective tissue disorders) | 27 | 37 | 53
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 15 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | 38 | 32
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 33 | 50 | 46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 37 | 45
Synovial cyst (Musculoskeletal and connective tissue disorders) | 6 | 12 | 17
Carpal tunnel syndrome (Nervous system disorders) | 8 | 12 | 20
Headache (Nervous system disorders) | 23 | 23 | 13
Hypoaesthesia (Nervous system disorders) | 22 | 42 | 50
Paraesthesia (Nervous system disorders) | 20 | 59 | 59
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 9

LIMITATIONS AND CAVEATS:
Due to FDA imposed clinical hold, enrollment was stopped prematurely and, therefore, not all study procedures and visits occurred as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.